CLINICAL TRIAL: NCT00106678
Title: Typology of Adherence in Adolescents: Phase II
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 023B
Record Dates: First submitted 2005-03-28; First posted 2005-03-29 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-02

CONDITIONS: HIV Infection
Keywords: HIV; Antiretroviral therapy (ART); HAART; Adherence; Barriers
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infected through risk behaviors
- Infected perinatally or through blood/blood products.

SUMMARY:
A number of factors influence HIV-positive adolescents' acceptance of and willingness to continue taking anti-HIV medicines. These factors include mental health and substance abuse issues, barriers such as lack of medical insurance, and cognitive-behavioral barriers (such as a person's impression of the impact of the medicines on his/her health and a person's sense of his/her ability to continue taking the medications prescribed). The purpose of this study is to use a survey to determine how common specific barriers are that prevent HIV positive adolescents from taking their anti-HIV medicines and if those barriers cluster together. The information collected will be used to develop and validate a schema for classifying HIV medication adherence by barriers to adherence or clusters of barriers to adherence. This classification schema could then be used in the development of interventions that better meet the needs of HIV-infected youth.

DETAILED DESCRIPTION:
As more HIV-infected adolescents are identified and linked into care, the dyad of medication and medication adherence continues to be an issue for both the provider and the patients. Thus, developing a strategy to assess adherence and barriers to adherence in this population is integral so that interventions can be targeted towards adolescents' specific needs. Our operating premise is that the issue of drug adherence is multi-factorial and that interventions that combine a variety of modalities may be preferred. However, before such interventions can be developed, we must first develop a tool that can be used to assess medication adherence and to identify barriers to medication adherence in this population.

This is a cross-sectional survey designed to assess the most prevalent combination of barriers to HIV medication adherence in adolescents. Specific barriers focused on in this study include mental health disorders, substance abuse, and cognitive-behavioral and structural barriers. In this Phase II study, the Adherence Staging Algorithm and the Participant Assessment Tool, pilot tested and modified based on findings from Phase I of the study, will be used to determine the prevalence of the specific barriers to adherence among HIV-infected youth requiring antiretroviral medication and the most common clusters of specific barriers. A cognitive-behavioral barriers schema for classifying HIV medication adherence in adolescents will be developed and validated.

The study consists of a one-time visit with a face-to-face interview to complete two questionnaires: the Adherence Staging Algorithm to classify the subject's adherence to his/her prescribed medications, and the Participant Assessment Tool to assess the prevalence of barriers to adherence that the subjects may have experienced. The interview takes no more than 30 minutes. In addition, the patient's medical record will be reviewed for HIV-related clinical data such as viral load, CD4, history of medications prescribed, and barriers the patient may have experienced such as mental health or substance abuse problems.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 12 years and 24 years
* Eligible for ART (antiretroviral therapy) based on US Public Health Service guidelines
* Have been offered and/or prescribed HAART (highly active antiretroviral therapy)
* Ability to give informed consent or assent with parental permission, where required

Exclusion Criteria:

* Infected with HIV but do not require ART
* Started HAART but stopped due to medical reasons, (e.g., change in medication guidelines, toxicity, resistance, etc.)
* Females prescribed/receiving HAART for the purpose of preventing mother-to-child transmission

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of HIV-infected youth who are eligible for antiretroviral therapy (ART) based on the US Public Health Service (PHS) guidelines and have been offered and/or prescribed HAART by their healthcare provider. Subjects aged 12 through 24 years old will be recruited from youth engaged in care at the fifteen ATN clinical sites located across the United States and in Puerto Rico. Youth engaged in care at selected non- ATN clinic centers will also be offered the opportunity to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2004-06; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Rudy, MD, Study Chair — Children's Hospital of Philadelphia
Locations (17):
- United States (16):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane University, New Orleans, Louisiana
  - University of Maryland Medical School, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Childrens Hospital Boston, Boston, Massachusetts
  - Weill Medical College of Cornell University-New York Presbyterian Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- University Pediatric Hospital, San Juan, Puerto Rico